CLINICAL TRIAL: NCT06691035
Title: Immunologic Targeting of Native and Mutated ESR1 Receptor for Treatment of Hormone Receptor Expressing Metastatic Breast Cancer
Brief Title: Immunologic Targeting of ESR1 Receptor for Hormone Receptor Expressing Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: The V Foundation for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-23161
Record Dates: First submitted 2024-11-14; First posted 2024-11-15 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer Metastatic Breast Cancer; HER2-negative Breast Cancer
Keywords: HER-2 Negative Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — elacestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Elacestrant + DC1 (Experimental): Patients will undergo apheresis of peripheral blood to collect and create DC1 vaccines. DC1 will be pulsed with ESR1 native or mutated peptides. After DC1 vaccines have undergone safety testing and are ready to be used, patients will be injected in groin nodes (or accessible breast tumor if available) weekly with these pulsed DC1 for eight consecutive weeks. They will alternate between native ESR1 DC1s and mutated ESR1 DC1s.
  Patients will receive combination of DC1 vaccinations and Elacestrant concurrently.
  Elacestrant is a novel oral selective estrogen downregulator, administered during vaccination and continued after.
  Elacestrant is considered standard of care for patients with ESR1 mutated HR+ HER2-metastatic breast cancer.
  Pulsed DC1 will be administered after initial induction every four weeks x 3 doses.
  Interventions: Drug: Elacestrant; Biological: DC1 native/mutated ESR1

INTERVENTIONS:
Drug: Elacestrant — 345 mg (or 86 mg tablets) orally daily during vaccination and continued after until progression.
  Cycle Length 28 days (4 weeks)
  Other Names: Oserdu
Biological: DC1 native/mutated ESR1 — 2.0-5.0 x 10 (20-50 million) cells (Injections in groin nodes (or accessible breast tumor if available) weekly with DC1 for eight consecutive weeks, alternating between native ESR1 DC1s and mutated ESR1 DC1s.
  Mutated ESR1 DC1s on week 1 followed by native ESR1 DC1s on week 2, alternating during the initial vaccination series and the subsequent booster phase.
  Pulsed DC1 will be administered after initial induction every four weeks x 3 doses.

SUMMARY:
This is a pilot study to determine feasibility and safety of the combination of Dendritic Cell (DC1) vaccines and elacestrant in patients with hormone positive HER2 negative metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed diagnosis of hormone positive HER2 negative metastatic breast cancer per ASCO/CAP criteria, with diagnosis established through either a breast/axillary biopsy or biopsy of a metastatic lesion.

  1. Estrogen Receptor (ER) or Progesterone Receptor (PR) are considered positive when expressed ≥1% on immunohistochemistry (IHC).
  2. HER2 is considered negative by IHC when expression is 0 or 1+ and if equivocal 2+ then a reflex in situ hybridization should be not amplified (standard practice per ASCO/CAP criteria).
* Participants must have Presence of an ESR1 mutation detected via tissue based or blood based (ctDNA) genomic profiling.
* Participants must have been previously treated with at least 1 line of endocrine therapy and a CDK 4/6 inhibitor in the metastatic setting.
* Participants must have measurable or nonmeasurable (evaluable) disease on imaging by RECIST v1.1.
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
* Participants must be adults 18 years or older.
* Participants must have the ability to understand and the willingness to sign a written informed consent document.
* Participants must be able to read and speak standard English or Spanish.
* Participants must have adequate organ and marrow function as defined below:

  1. absolute neutrophil count ≥1,000/mcL
  2. platelets ≥75,000/mcL

  d. AST(SGOT)/ALT(SGPT) ≤3 fold × institutional ULN e. creatinine 1.5 ≤ institutional ULN f. hemoglobin (Hb) ≥ 9 g/dL g. Total bilirubin < 1.5 x ULN or <3 x ULN in the presence of documented Gilbert's syndrome unconjugated hyperbilirubinemia)
* Participants must have a negative pregnancy test for pre-menopausal women of childbearing potential.
* Participants that are pre-menopausal women of childbearing potential who are sexually active with a male partner must agree to use adequate contraception prior to the study, for the duration of study participation.
* Inclusion of minorities: patients of all races and ethnic groups who meet the above inclusion and below exclusion criteria are eligible for this trial.
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Participants must have the ability to understand and the willingness to sign a written informed consent document or have a legally authorized representative sign on the participant's behalf.
* Participants with treated and stable brain metastases are eligible if brain imaging shows no evidence of progression within 2 months of trial enrollment.

Exclusion Criteria:

* Pregnant women are excluded from this study because study treatment agent(s) used in this study may have the potential for teratogenic or abortifacient effects. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with agents used in this study, breastfeeding should be discontinued if the mother is treated with study agents used in this study.
* Previous treatment with Elacestrant.
* History of allergic reactions attributed to the study drugs.
* Active, progressing or newly diagnosed CNS metastases, including leptomeningeal carcinomatosis, because systemic treatment would need to be paused for these patients.
* Treatment with any investigational compound within 21 days prior to the first dose of study drugs or during this study.
* 14 day washout periods from previous anticancer therapy(ies) is required prior to enrollment including:

  * Cytotoxic chemotherapy
  * Tamoxifen or aromatase inhibitors
  * Fulvestrant
  * Targeted agents such as CDK 4/6 inhibitors, PIK3CA inhibitors, MTOR inhibitors
* Diagnosis or treatment for another systemic malignancy within 2 years before the first dose of study drugs, or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Uncontrolled intercurrent illness including-but not limited to-ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with advanced, symptomatic visceral spread, that are at risk of life-threatening complications in the short term, including massive uncontrolled effusions (peritoneal, pleural, pericardial), pulmonary lymphangitis.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome.
* Active infection including tuberculosis, hepatitis B (known positive HBV surface antigen [HbsAg]), or hepatitis C (HCV). Participants with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HbsAg) are eligible. Participants with positive Hepatitis C Virus (HCV) antibody are eligible if polymerase chain reaction is negative for HCV RNA.
* Concurrent or prior use of immunosuppressive medication within 14 days before the first dose of study drugs, with the following exceptions: premedication with dexamethasone, intranasal, inhaled, topical or local steroid injections, systemic corticosteroids at physiologic doses not exceeding 10 mg/day of prednisone or its equivalent; steroids as premedication for hypersensitivity reactions (e.g., premedication for iodinated contrast allergy before CT scan).
* Inability to comply with protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Rate of Successful Completion | Up to 2 years
  Feasibility: Defined as a patient's ability and willingness to complete the treatment regimen (8 weeks) to End of Treatment (EOT) (window of + 30 days from date of last study treatment).
  Data collection will include rate of successful completion.
Occurrence Rate | Up to 2 years
  Feasibility: Defined as a patient's ability and willingness to complete the treatment regimen (8 weeks) to End of Treatment (EOT) (window of + 30 days from date of last study treatment).
  Data collection will include occurrence rate for each reason stated for non-completion.
Occurrence of Treatment Related Adverse Events | Up to 2 years
  Number of participants with treatment related adverse events, per event category.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 2 years
  Progression Free Survival (PFS) is measured from the start of treatment until disease progression or death from any cause.
Clinical Benefit Rate (CBR) | Up to 2 years
  Clinical Benefit Rate (CBR) is measured by Complete Response (CR) + Partial Response (PR) + Stable Disease.
Overall Response Rate (ORR) | Up to 2 years
  Overall Response Rate (ORR) is measured by Complete Response (CR) + Partial Response (PR).

OTHER OUTCOMES:
Dose Limiting Toxicity | Up to 2 years
  Dose limiting toxicity (DLT) is defined as grade ≥ 3 non-hematologic toxicity; grade ≥ 3 hematologic toxicity thought be at least possibly related to vaccines.
  Toxicity data will be reviewed after small groups of patients have been treated and observed for 30 days after the last vaccination.
  The study will enroll a total number of 18 patients. Enrollment will be suspended if data suggest that the rate of unacceptable vaccine-related toxicity exceeds 25%.

CONTACTS AND LOCATIONS:
Overall Officials: Aixa Soyano Muller, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — http://www.moffitt.org/clinical-trials-research/clinical-trials/